CLINICAL TRIAL: NCT02775708
Title: Development of Applications of the ® PillCam Endoscopy System and Evaluation of Their Performance
Acronym: NOISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COVGIRD0477
Record Dates: First submitted 2016-04-20; First posted 2016-05-18 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-09

CONDITIONS: Any Gastric Condition Which Requires Capsule Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsule endoscopy (Experimental): open label arm ; up to 100 subjects indicated for capsule endoscopy (CE) procedure will undergo the CE procedure with the Pillcam endoscopy system
  Interventions: Device: Pillcam endoscopy system

INTERVENTIONS:
Device: Pillcam endoscopy system

SUMMARY:
The purpose of this study is to support development of PillCam Endoscopy System applications.

ELIGIBILITY:
Inclusion Criteria:

* Subject's from 18 years of age.
* Subject is indicated for Capsule Endoscopy procedure.
* Subject agrees to sign the Informed Consent Form.

Exclusion Criteria:

* Female subject is pregnant.
* Subject is known or is suspected to suffer from intestinal obstruction (symptoms such as severe abdominal pain with accompanying nausea or vomiting).
* Subject has a pacemaker or other implanted electro-medical device.
* Subject has any condition, which precludes compliance with study and/or device instructions, such as swallowing problems.
* Subject suffers from life threatening conditions.
* Subject is currently participating in another clinical study that may directly or indirectly affect the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Number of gaps in the RAPID video will be assessed | capsule endoscopy procedure day

CONTACTS AND LOCATIONS:
Locations (2):
- Klinikum Furth, Fürth, Germany
- Hospital De Navarra, Pamplona, Navarre, Spain